CLINICAL TRIAL: NCT07357935
Title: Early Inflammatory-Immune Stratification and Precision Glucocorticoid Intervention in Acute Respiratory Failure Induced by Community-Acquired Pneumonia
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qingyuan Zhan (Other)
Collaborators: The First Affiliated Hospital of Guangzhou Medical University (Other); Wuhan Metware Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor-Investigator, Qingyuan Zhan, Director, China-Japan Friendship Hospital
Organization: China-Japan Friendship Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZD01902401
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure; Community-Acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — Methylprednisolone; Methylprednisolone Hemisuccinate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standardized Methylprednisolone Intervention (Dose-Adjusted) (Experimental): All enrolled patients receive intravenous methylprednisolone (0.5-1 mg/kg/day, dissolved in 100ml normal saline, once daily) for a total of 7 days. The initial dose is determined by the oxygenation index (PFR) at enrollment:
  * PFR ≤ 150 mmHg: Methylprednisolone 1 mg/kg/day.
  * PFR > 150 mmHg: Methylprednisolone 0.5 mg/kg/day.
  At day 4 (D4), the dose is halved if the patient shows a clinical response (defined as an improvement in the oxygenation index ≥20% AND a decrease in SOFA score ≥2 points); otherwise, the original dose is maintained. Methylprednisolone is discontinued upon death or transfer out of the ICU. All patients also receive standard care for bacterial CAP-ARF as determined by the treating physician.
  Interventions: Drug: Methylprednisolone

INTERVENTIONS:
Drug: Methylprednisolone — This is the core intervention. For detailed dosage, administration, and dose-adjustment strategy, please refer to the Arm Description.
  Other Names: Solu-Medrol

SUMMARY:
This is a prospective, multicenter, interventional cohort study aimed at constructing a high-quality, dynamic multimodal database for patients with acute respiratory failure caused by community-acquired pneumonia (CAP-ARF). The study focuses on bacterial CAP-ARF patients receiving standardized glucocorticoid therapy to investigate the heterogeneity of treatment responses under different etiologies and immune statuses. The goal is to provide a data foundation for precise immune stratification and identification of glucocorticoid-sensitive populations.

DETAILED DESCRIPTION:
This study is part of the National Major Science and Technology Project for the Prevention and Control of Emerging and Major Infectious Diseases. It integrates existing multicenter cohorts (including healthy individuals, non-infectious ARF, mild CAP, and CAP-ARF patients) and establishes a prospective, standardized glucocorticoid intervention cohort for bacterial CAP-ARF. Eligible patients (age ≥18, admitted to ICU ≤48 hours, meeting bacterial pneumonia and severe ARF criteria) are treated with methylprednisolone based on initial oxygenation index (PFR ≤150 mmHg: 1 mg/kg/d; PFR >150 mmHg: 0.5 mg/kg/d). Dosing is adjusted at day 4 based on clinical response (improvement in oxygenation and SOFA score), with a total treatment duration of 7 days. Multimodal data-including clinical information, inflammatory/immune biomarkers, chest CT imaging, and multi-omics sequencing (transcriptomics, proteomics, metabolomics)-are collected at multiple timepoints (baseline, day 4, day 8). The database will support the analysis of immune-inflammatory profiles, identification of glucocorticoid-responsive subgroups, and development of precision intervention strategies for CAP-ARF.

ELIGIBILITY:
Inclusion Criteria:1. Age ≥ 18 years. 2. Admitted to the Intensive Care Unit (ICU) within 48 hours. 3. Meet diagnostic criteria for bacterial community-acquired pneumonia (CAP). 4. Meet at least one severity criterion: a) Receiving mechanical ventilation for acute respiratory failure with PEEP ≥ 5 cmH2O; OR b) On high-flow oxygen with FiO2 ≥ 0.5 and PaO2/FiO2 ratio ≤ 250 mmHg; OR c) On a reservoir oxygen mask with PaO2 below the specified flow threshold (see protocol). 5. Signed informed consent.

-

Exclusion Criteria: 1. Suspected aspiration pneumonia. 2. Invasive mechanical ventilation within 14 days prior to admission. 3. Diagnosis of hospital-acquired or ventilator-associated pneumonia (HAP/VAP). 4. Positive for influenza virus, active tuberculosis, or fungal infection (except Pneumocystis jirovecii). 5. Active viral hepatitis or herpesvirus infection. 6. Hypersensitivity to glucocorticoids, or contraindications as judged by the investigator (e.g., severe concurrent infections, active gastrointestinal hemorrhage). 7. High-dose glucocorticoid therapy (>1 mg/kg/day prednisone equivalent) within 30 days for underlying disease. 8. Death within 24 hours of ICU admission. 9. Pregnancy or lactation. 10. Participation in other interventional studies or refusal to participate.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
90-day all-cause mortality | At Day 90 (from enrollment)
  The proportion of participants who die from any cause within 90 days after enrollment.
28-day all-cause mortality | : At Day 28 (from enrollment)
  The proportion of participants who die from any cause within 28 days after enrollment.

SECONDARY OUTCOMES:
Incidence of glucocorticoid-related adverse events (AEs) | From the first dose of methylprednisolone up to Day 28 (the end of the primary safety observation period).
  The occurrence of AEs known to be associated with glucocorticoid therapy, including but not limited to: secondary infection, hyperglycemia, myopathy/weakness, gastrointestinal bleeding, sodium/water retention, and inflammatory rebound.
Proportion of participants with glucocorticoid responsiveness at Day 4 | At Day 4 (from enrollment)
  The proportion of participants who meet the pre-defined criteria for glucocorticoid responsiveness at Day 4 (D4) after initiating treatment. Responsiveness is defined as: an improvement in the oxygenation index (PFR) by ≥20% AND a decrease in Sequential Organ Failure Assessment (SOFA) score by ≥2 points compared to baseline (D1).